CLINICAL TRIAL: NCT06671522
Title: In-depth Survey for the Reasons of Weight Control Difficulties
Acronym: Weight Control
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: O-BW-001
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Weight Control
Keywords: Deep survey of weight control difficulty
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obesity
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — It is a qualitatative research. Only a survey.

SUMMARY:
The aim of this study was to investigate the causes of weight control difficulties in overweight or obese patients .Overweight or obese Chinese patients were enrolled. According to their age, 3 males and 3 females (24 in total) aged 14-20 years, 21-40 years, 41-60 years and 61-80 years were included for interview for about 1 hour. The interview included demographic basic information and other characteristics, time and results of weight control, and causes of weight control difficulties. After collecting the information, classification and summary analysis were performed.

DETAILED DESCRIPTION:
The aim of this study was to investigate the causes of weight control difficulties in overweight or obese patients of all ages by in-depth interview, in order to explore more causes of weight control difficulties, to make early exploration for targeted large-scale cross-sectional survey studies on the causes of weight control difficulties in the future, and to find the causes of weight control difficulties, which will help to study measures to solve weight control difficulties.

Study design: Overweight or obese Chinese patients were enrolled. According to their age, 3 males and 3 females (24 in total) aged 14-20 years, 21-40 years, 41-60 years and 61-80 years were included for interview for about 1 hour. The interview included demographic basic information and other characteristics, time and results of weight control, and causes of weight control difficulties. After collecting the information, classification and summary analysis were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, nature and method of the study, voluntarily participate in the study, agree to record the interview content through a tape recorder during the interview, and sign the informed consent form (ICF) before the interview;
2. Chinese aged 14-80 years (including boundary value, subject to the time of signing the informed consent form), male or female;
3. Patients with body mass index (BMI) greater than 24 kg/m 2 , who have taken any weight control measures;
4. Willing and able to comply with study requirements. -

Exclusion Criteria:

1. Inability to communicate in speech; 2. Known mental or psychological disorder of any kind; 3. Other conditions that, in the opinion of the investigator, would make participation in this study inappropriate.

-

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight or obese Chinese patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reasons of weight control difficulty | Before the time of interview

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
There might be some individual data with sensitive, will decide after completion of the study.